CLINICAL TRIAL: NCT01221857
Title: Allogeneic Stem Cell Transplantation of NiCord®, Umbilical Cord Blood-Derived Ex Vivo Expanded Stem and Progenitor Cells, in Combination With a Second, Unmanipulated Cord Blood Unit in Patients With Hematological Malignancies
Brief Title: Pilot Study Evaluating Safety & Efficacy of DCBT: NiCord® & UNM CBU to Patients With Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC P#01.01.020
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Acute Myelogenous Leukemia (AML); Myelodysplastic Syndrome (MDS); Non-Hodgkin's Lymphoma; Hodgkin's Disease
Keywords: Double Umbilical Cord Blood Stem Cell Transplantation; Hematological Malignancies; HLA Mismatched Donors; Cord Blood Transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NiCord (Experimental)
  Interventions: Drug: NiCord®

INTERVENTIONS:
Drug: NiCord® — NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells.

SUMMARY:
Pilot Study Evaluating the Safety and Efficacy of a Co-Transplantation of NiCord®, a UCB-derived ex Vivo Expanded Population of Stem and Progenitor Cells with a Second, Unmanipulated CBU in Patients with Hematological Malignancies

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) is a potentially curative procedure for various hematological malignancies, bone marrow failure syndromes and inherited metabolic disorders. The application of allogeneic HSCT is limited by donor availability such that only approximately one-third of the otherwise appropriate candidates have suitably matched family donors. Alternative donors include mismatched family members or matched unrelated donors, but these approaches are often complicated by an increased risk of graft-versus-host disease (GvHD) and a prolonged and cumbersome search and procurement process. In addition, far fewer subjects of racial minorities find suitable human leukocyte antigen (HLA)-matched donors.

Umbilical cord blood has been increasingly used as an alternative source of stem cells and has extended the availability of allogeneic HSCT to patients who would otherwise not be eligible for this curative approach. In the last decade the number of cord blood transplantations from related and unrelated donors has increased dramatically. It is estimated that more than 20,000 patients have undergone cord blood transplantation from unrelated donors to date for a variety of genetic, hematological, immunological, metabolic and oncologic disorders. The major advantages of cord blood transplantation include easy procurement, no risk to donors, reduced incidence of transmitting infections, immediate availability, and reduced risk of acute GvHD in the setting of donor-recipient HLA mismatch. Nevertheless, the low cell dose remains a main limitation of this cell source leading to delayed hematopoietic reconstitution, higher risk of graft failure and relatively high treatment related mortality rates as compared to other hematopoeitic cell sources. To improve outcomes and extend applicability of cord blood transplantation, one potential solution is ex vivo expansion of cord blood-derived stem and progenitor cells.

The Sponsor has undertaken to develop NiCord®, which is based on a novel technology for ex vivo cell expansion of cord blood derived hematopoietic progenitor cells. By increasing the number of the short and long-term reconstitution progenitor cells transplanted, NiCord® has the potential to enable broader application of umbilical cord blood transplantation and improve clinical outcomes in subjects with high-risk hematological malignancies.

The main objective of the current study is to evaluate the safety of co-transplantation of NiCord® and an unmanipulated cord blood unit in patients with hematological malignancies following myeloablative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Applicable disease and eligible for myeloablative SCT
* Patients must have two partially HLA-matched CBUs
* Back-up stem cell source
* Adequate Karnofsky Performance score or Lansky Play-Performance scale
* Sufficient physiological reserves
* Signed written informed consent

Exclusion Criteria:

* HLA-matched related donor able to donate
* Prior allogeneic HSCT
* Lymphoma patients with progressive disease
* Other active malignancy
* Human immunodeficiency virus (HIV) infection
* Active or uncontrolled infection
* Active/symptoms of central nervous system (CNS) disease
* Pregnancy or lactation

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Snyder, PhD, Study Director — Gamida Cell ltd; Joanne Kurtzberg, MD, Principal Investigator — Duke University; Mitchell Horwitz, MD, Principal Investigator — Duke University; Patrick Stiff, MD, Principal Investigator — Loyola University
Locations (2):
- United States (2):
  - Loyola University, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Horwitz ME, Chao NJ, Rizzieri DA, Long GD, Sullivan KM, Gasparetto C, Chute JP, Morris A, McDonald C, Waters-Pick B, Stiff P, Wease S, Peled A, Snyder D, Cohen EG, Shoham H, Landau E, Friend E, Peleg I, Aschengrau D, Yackoubov D, Kurtzberg J, Peled T. Umbilical cord blood expansion with nicotinamide provides long-term multilineage engraftment. J Clin Invest. 2014 Jul;124(7):3121-8. doi: 10.1172/JCI74556. Epub 2014 Jun 9. PMID 24911148
- [Derived] Peled T, Shoham H, Aschengrau D, Yackoubov D, Frei G, Rosenheimer G N, Lerrer B, Cohen HY, Nagler A, Fibach E, Peled A. Nicotinamide, a SIRT1 inhibitor, inhibits differentiation and facilitates expansion of hematopoietic progenitor cells with enhanced bone marrow homing and engraftment. Exp Hematol. 2012 Apr;40(4):342-55.e1. doi: 10.1016/j.exphem.2011.12.005. Epub 2011 Dec 20. PMID 22198152
- See also: Gamida Cell Ltd. — http://www.gamida-cell.com
- See also: Duke University Medical Center — http://www.dukehealth.org
- See also: Loyola University — http://www.loyolamedicine.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 patients were enrolled/transplanted; efficacy results were summarized for 11 patients treated with NiCord. 1 patient was transplanted with unmanipulated cord only. Safety results were summarized for all patients.
Groups:
- NiCord: NiCord: NiCord is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells.
Period: Overall Study
Arm/Group | NiCord
Started | 12
Completed (1 patient received unmanipulated cord only.) | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NiCord
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 45 [21 to 61]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Acute Toxicity Associated With the Infusion of NiCord
Description: Acute toxicity associated with the infusion of NiCord will be measured by adverse events within 24 hours post-infusion, defined as the acute toxicity period. Known adverse events associated with myeloablation and cord blood transplant were specifically monitored including fever, chills, allergic reaction/hypersensitivity, anaphylaxis, sinus bradycardia, sinus tachycardia, hypertension, hypotension, nausea, vomiting, diarrhea, dyspnea, hypoxia, hemoglobinuria, infection, flank pain and any other skin, CNS, cardiac, pulmonary or other toxicity manifestations.
Time Frame: 180 days post-transplant
Population: Patients transplanted with NiCord
Measure: Count of Participants; unit: Participants
Groups:
- NiCord: Analysis population is patients transplanted with NiCord plus unmanipulated cord blood unit.
Arm/Group | NiCord
Number analyzed (Participants) | 11
Participants | 0

2. Primary Outcome: Proportion of Patients With Neutrophil Engraftment
Description: Neutrophil engraftment was defined as achieving an Absolute Neutrophil Count (ANC) of ≥500 mm3 for 3 consecutive measurements on different days by day 42 inclusive (the day of engraftment was defined as the first of these 3 days). The ANC recovery must be of donor origin documented by peripheral blood chimerism assays indicating less than or equal to 10% host cells in peripheral blood.
Time Frame: 42 days
Population: Patients transplanted with NiCord
Measure: Number; unit: proportion of patients
Groups:
- Neutrophil Engraftment: Patients transplanted with NiCord plus unmanipulated cord blood unit.
Arm/Group | Neutrophil Engraftment
Number analyzed (Participants) | 11
proportion of patients | 0.91

3. Secondary Outcome: Proportion of Patients Who Developed Acute GvHD Grade II-IV and III-IV
Description: Acute GvHD was assessed from transplantation (day 0) until day 99 post-transplant or more frequently as clinically indicated. GvHD was classified according to the Glucksberg Classification (Glucksberg, Storb et al. 1974).
  The overall grade of GvHD, however, was determined by an assessment of skin disease, liver disease and gastrointestinal manifestations.
Time Frame: 180 days
Measure: Number; unit: proportion of patients
Groups:
- Grade II-IV GvHD: All patients transplanted were assessed for acute GvHD grade II-IV.
- Grade III-IV GvHD: All patients transplanted were assessed for acute GvHD grade III-IV.
Arm/Group | Grade II-IV GvHD | Grade III-IV GvHD
Number analyzed (Participants) | 11 | 11
proportion of patients | 0.45 | 0

4. Secondary Outcome: Non-relapse Mortality
Description: Proportion of patients who had non-relapse mortality at 100 days.
Time Frame: 100 days
Measure: Number; unit: proportion of patients
Groups:
- Non-relapse Mortality: proportion of patients with non-relapse mortality at 100 days
Arm/Group | Non-relapse Mortality
Number analyzed (Participants) | 11
proportion of patients | 0.09

ADVERSE EVENTS:
Arm/Group | NiCord
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NiCord (N=12)
Pneumonia (Infections and infestations) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Altered mental status (Psychiatric disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Graft rejection (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Disease relapse (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NiCord (N=12)
Hypertension (Cardiac disorders) | 6 (7)
Hypomagnesemia (Investigations) | 4 (4)
aGvHD (Immune system disorders) | 7 (10)
CMV reactivation (Infections and infestations) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4)
Hypotension (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3)
HHV-6 Reactivation (Infections and infestations) | 6 (6)
Staph Coagulase Infection (Infections and infestations) | 2 (3)
Hypocalcemia (Investigations) | 3 (3)
BK virus infection (Infections and infestations) | 2 (2)
Elevated LFTs (Gastrointestinal disorders) | 1 (1)
E coli infection (Infections and infestations) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
RSV infection (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Enterococcus infection (Infections and infestations) | 1 (1)
CMV gastritis (Gastrointestinal disorders) | 1 (1)
Hypoalbuminemia (Investigations) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No